CLINICAL TRIAL: NCT06111534
Title: Paternal vs Maternal Holding-Cuddling for Procedural Pain in Healthy Term Neonates: A Quasi-experimental Study
Brief Title: Paternal vs Maternal Holding-Cuddling for Procedural Pain in Healthy Term Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2016/13173
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Procedural Pain
Keywords: Healthy infant; Parent participation; Procedural pain
MeSH Terms: conditions — Pain, Procedural

STUDY DESIGN:
Intervention Model Description: Participants were recruited using random sampling. The group assignment was determined using the closed envelope method. Therefore, data were collected first from the MHC group, followed by the PHC and control groups.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MHC group (Experimental): Each MHC group participant (n=30) was brought to the procedure room by its mother. The mother sat in a comfortable chair with back support. She held her baby close to her chest, with the baby's head in a crossed position so that it could see its mother. The same nurse collected the blood sample. The mother communicated with the baby verbally and made eye contact with it to calm it down during the procedure. She was holding the baby both during and after the procedure.
  Interventions: Behavioral: Holding
- PHC group (Experimental): Each PHC group participant (n=30) was brought to the procedure room by its father. The father sat in a comfortable chair with back support. He held his baby close to his chest, with the baby's head in a crossed position so that it could see its father. The same nurse collected the blood sample. The father communicated with the baby verbally and made eye contact with it to calm it down during the procedure. He was holding the baby both during and after the procedure.
  Interventions: Behavioral: Holding
- Control group (No Intervention): The control group participants (n=32) underwent the procedure according to the routine clinical practice. Either parent brought the baby into the procedure room and laid it on the procedure table in the supine position. The nurse collected the blood sample. The parent was present in the room and communicated with the baby only verbally during the procedure. The parent picked up the baby after the procedure.

INTERVENTIONS:
Behavioral: Holding — Holding is an effective non-pharmacological method for reducing procedural pain. Minor painful procedures, such as heel pricks, are easy to use, practical, non-invasive, and affordable procedures when performed when the neonate is held/cuddled by one of its parents. Neonates held/cuddled by their mothers are likely to experience less pain and cry less during heel pricks. The MHC and PHC methods help neonates experience tactile, auditory, visual, and olfactory sensory inputs that can enhance analgesic effects. These multisensory methods can alleviate the pain experienced by the infant during minor painful procedures and shorten the crying time. This type of analgesia may be mediated by multisensory stimulation associated with the mother/father-infant attachment.
  Arms: MHC group; PHC group

SUMMARY:
This study investigated the effect of maternal holding-cuddling (MHC) and paternal holding-cuddling (PHC) on heel prick pain and crying duration in healthy term neonates

DETAILED DESCRIPTION:
Newborns undergo many painful procedures. The heel prick, or heel lancing, is a painful procedure used for newborn screening tests. It is a more painful procedure than other venipuncture procedures. All pediatricians and healthcare professionals working with neonates should focus on pain management during heel pricks for two reasons. First, they are under an ethical obligation to help neonates experience as little pain as possible during medical procedures. Second, repeated painful exposure has harmful consequences. The International Guide to Pediatric Anesthesia (Good Practice in Postoperative and Procedural Pain) also recommends pharmacological and non-pharmacological methods to prevent and effectively manage acute procedural pain in children. However, pharmacological methods for pain management in neonates may have some side effects. On the other hand, non-pharmacological methods are easy to use, affordable, and time-effective methods with no side effects. Healthcare professionals do not use non-pharmacological methods that are expensive, hard to apply, and time-consuming. Therefore, this study focused on maternal holding-cuddling and paternal holding-cuddling as alternative non-pharmacological methods to prevent procedural pain in neonates during heel pricks. Holding-cuddling is an effective non-pharmacological method for reducing procedural pain.

ELIGIBILITY:
Inclusion Criteria:

* healthy term neonates
* birth weight between 2500 and 4000 g
* 38-42 gestational week
* postnatal age of 48-72 hours
* a 5-minute APGAR score of ≥8,
* having had no experience of any painful interventions other than vitamin K and hepatitis B vaccine at birth
* fed between 30 and 60 min before the procedure
* undergoing heel prick only once
* blood collection for the Guthrie test
* willing to hold their babies during the procedure

Exclusion Criteria:

* sleeping during the procedure
* receiving analgesics up to 24 hours before the procedure

Ages: 38 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 92 (Actual)
Dates: Start 2016-02-04 (Actual); Primary Completion 2016-08-20 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Neonatal Infant Pain Scale (NIPS) | Through painful procedure completion, an average of 10 minutes
  The scale is used to assess procedural pain in neonates. It is a behavioral scale assessing five behavioral indicators (facial expression, cry, arms, legs, and state of alertness) and one physiological indicator (breathing patterns). Five items (facial expression, breathing pattern, arms, legs, and state of alertness) are scored as 0 (Good) or 1 (Bad), while one item (crying) is scored as 0 (Good), 1, or 2 (Bad). The total scale score ranges from 0 to 7, with higher scores indicating more pain.

SECONDARY OUTCOMES:
Crying time during the procedure | Through painful procedure completion, an average of 2 minutes
  The duration of total crying time during the procedure is between when the heel is pricked and the injection site is covered with a cotton pad.
Crying time after the procedure | Through painful procedure completion, an average of 2 minutes
  The total crying time after the procedure is between when the procedure is completed and the baby calms down.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Özdemir, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Kadıköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared after the article is published.

REFERENCES:
- [Background] Perry M, Tan Z, Chen J, Weidig T, Xu W, Cong XS. Neonatal Pain: Perceptions and Current Practice. Crit Care Nurs Clin North Am. 2018 Dec;30(4):549-561. doi: 10.1016/j.cnc.2018.07.013. PMID 30447813
- [Background] Dur S, Caglar S, Yildiz NU, Dogan P, Guney Varal I. The effect of Yakson and Gentle Human Touch methods on pain and physiological parameters in preterm infants during heel lancing. Intensive Crit Care Nurs. 2020 Dec;61:102886. doi: 10.1016/j.iccn.2020.102886. Epub 2020 Jun 27. PMID 32601011
- [Background] Johnston CC, Campbell-Yeo M, Filion F. Paternal vs maternal kangaroo care for procedural pain in preterm neonates: a randomized crossover trial. Arch Pediatr Adolesc Med. 2011 Sep;165(9):792-6. doi: 10.1001/archpediatrics.2011.130. PMID 21893645
- [Background] Lawrence J, Alcock D, McGrath P, Kay J, MacMurray SB, Dulberg C. The development of a tool to assess neonatal pain. Neonatal Netw. 1993 Sep;12(6):59-66. PMID 8413140
- [Background] Kucukoglu S, Aytekin A, Celebioglu A, Celebi A, Caner I, Maden R. Effect of White Noise in Relieving Vaccination Pain in Premature Infants. Pain Manag Nurs. 2016 Dec;17(6):392-400. doi: 10.1016/j.pmn.2016.08.006. Epub 2016 Oct 15. PMID 27751753